CLINICAL TRIAL: NCT05228002
Title: sFlt-1/PlGF Ratio: Impact on the Management of Patients With Suspected Pre-eclampsia
Acronym: PROSPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-AOI-02
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator): The monitoring criteria used will be the same as those usually used at the Nice University Hospital, according to the protocol of the department.
  For patients in the "standard" group, the biomarker results will be masked and then revealed afterwards for statistical analysis.
  Interventions: Other: sFlt-1/PlGF ratio - Active Comparator: Standard
- Biomarkers (Experimental): The monitoring decision will be made based on the ratio calculation:
  Ratio < 38: "Classic" monitoring with one prenatal visit per month 38 ≤ Ratio ≤ 85: Close outpatient monitoring Ratio > 85: Inpatient monitoring in Pathological Pregnancy
  Interventions: Other: sFlt-1/PlGF ratio - Experimental: Biomarkers

INTERVENTIONS:
Other: sFlt-1/PlGF ratio - Active Comparator: Standard — Blood test for biomarkers (sFlt-1/PlGF ratio) For patients in the "standard" group, the biomarker results will be masked and then revealed afterwards for statistical analysis.
  For the "biomarkers" group, the monitoring decision will be made based on the ratio calculation
  Arms: Standard
Other: sFlt-1/PlGF ratio - Experimental: Biomarkers — Blood test for biomarkers (sFlt-1/PlGF ratio) For patients in the "standard" group, the biomarker results will be masked and then revealed afterwards for statistical analysis.
  For the "biomarkers" group, the monitoring decision will be made based on the ratio calculation.
  Arms: Biomarkers

SUMMARY:
Pre-eclampsia is a specific pathology of pregnancy classically associating arterial hypertension with proteinuria. Its prevalence in industrialized countries is 3 to 8% of pregnancies, which makes it a frequent pathology, and it is responsible for 30% of premature deliveries. The consequences of this pathology can be very serious for the mother:renal insufficiency, hepatic cytolysis, retro-capsular hematoma of the liver, convulsions, disseminated intravascular coagulation. Moreover, the consequences on the fetus and the pregnancy are just as serious: intrauterine growth retardation, induced prematurity, retroplacental hematoma, fetal death in utero.

Pre-eclampsia therefore remains difficult to diagnose and to prognose. The diagnosis of pre-eclampsia based on blood pressure and proteinuria has a predictive value of 30% for adverse outcomes related to pre-eclampsia.

In recent years, new biomarkers have been studied: PlGF, a placental growth factor, and sFlt-1, the free fraction of its membrane receptor.The pathophysiology and specificity of these biomarkers, but especially their ratio, has been widely studied and demonstrated in the diagnosis and prognosis of preeclampsia.

Nevertheless, few studies have analyzed the impact of this report on the hospitalization of patients, except mainly a German study which showed a change in the decision to hospitalize in 16.9% of cases. On the other hand, no French study has been carried out on this subject. Finally, no professional recommendation fully integrates or clearly frames the use of the ratio in current practice. Its use therefore remains disparate between countries, but also within the same country, as in France, where few centers use it.

The decision to hospitalize a patient with suspected preeclampsia depends on the organization of the health care system. It therefore seems interesting to analyze the precise impact on hospitalizations of the use of a diagnostic and prognostic tool such as the sFlt-1/PlGF ratio with the specificities of the French health system, which favors outpatient management.The study would evaluate the use of this promising tool in the daily management of parturients, paving the way for the development of simple recommendations applicable in the various French maternity hospitals.

The hypothesis is that the use of the sFlt-1/PlGF ratio in patients with suspected pre-eclampsia would reduce the rate of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patient
* Affiliated to the Social Security
* Signature of informed consent
* Term > 24 week of amenorrhea and < 37 week of amenorrhea
* Single criterion among the following: (only one box below must be ticked to allow inclusion):

  * de novo hypertension (PAS ≥ 140 mmHg and/or PAD ≥ 90 mmHg) ;
  * worsening of pre-existing hypertension >10 mmHg (on PAS or PAD ) ;
  * worsening of pre-existing proteinuria;
  * Excessive edema AND significant weight gain (minimum 2kg/week);
  * Headache AND another clinical sign (edema, rapid weight gain);
  * Visual disturbances (phosphenes and/or visual blur) AND/OR tinnitus;
  * Sudden weight gain (> 1kg/week during the 3rd trimester);
  * Low platelet count (thrombocytopenia < 150 G/L);
  * Hepatic cytolysis (ASAT and/or ALAT > 2N) without associated pruritus or jaundice;
  * Suspicion of intrauterine growth retardation on obstetric ultrasound, with no other cause found (no hypertension or proteinuria, no clinical or biological signs of pre-eclampsia) and no abnormal fetal dopplers.

Exclusion Criteria:

* Minor patient
* Patient with poor clinical tolerance of hypertension and/or need for immediate introduction of intravenous antihypertensive therapy
* Patient with a specific complication of pre-eclampsia requiring immediate management at the time of inclusion: in utero fetal death, retroplacental hematoma, disseminated intravascular coagulation or emergency cesarean section.
* Association of at least 2 of the following criteria:

  * De novo proteinuria (24h proteinuria ≥ 0.3 g/24h or P/C ratio ≥ 0.3) or worsening of pre- existing proteinuria;
  * Criteria for clinical suspicion of pre-eclampsia: epigastric pain, excessive edema, headaches, visual disturbances, sudden weight gain (> 1kg/week in the 3rd trimester);
  * Biological signs associated with pre-eclampsia: low platelet count (thrombocytopenia < 150 G/L), hepatic cytolysis (ASAT and/or ALAT > 2N);
  * Suspicion of intrauterine growth retardation on obstetrical ultrasound, with no other cause found.

A combination of at least 2 of these criteria raises the suspicion of pre-eclampsia, and, according to the new CNGOF recommendations of 2024, requires systematic initial hospitalization.

- Vulnerable person requiring enhanced protection, i.e., relatively (or totally) unable to protect their own interests. Specifically, the person's power, intelligence, education, resources, strength, or other attributes necessary to protect his or her own interests may be inadequate (e.g., persons deprived of liberty, minors, persons under guardianship, persons with mental or emotional disabilities in the broadest sense of the word, illiterate persons, refugees and asylum seekers, alcoholics and drug addicts, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 43 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
hospitalization rate | up to 4 months
  hospitalization rate for each group.

SECONDARY OUTCOMES:
sFlt-1/PlGF ratio at inclusion and length of hospital stay | up to 4 months
  correlation between sFlt-1/PlGF ratio at inclusion and length of hospital stay
Complications specific to pre-eclampsia | up to 4 months
  occurrence of complications specific to pre-eclampsia (eclampsia, HELLP-syndrome, fetal death in utero...)
Pregnancy Outcome | up to 4 months
  Correlation of the sFlt-1/PlGF ratio at inclusion and its kinetics with pregnancy outcome (route of delivery and urgency criteria)
newborn health status at birth | up to 4 months
  Correlation of the sFlt-1/PlGF ratio at inclusion and its kinetics with newborn health status at birth (Apgar score and need for immediate pediatric management)

CONTACTS AND LOCATIONS:
Overall Officials: Julie ANTOMARCHI, Principal Investigator — Nice University Hospital
Locations (1):
- Nice University Hospital, Nice, France